CLINICAL TRIAL: NCT05853289
Title: Piloting a Web-Based Implementation Resource for Pregnancy Opioid Use Disorder Care in Jail
Brief Title: Piloting a Web Resource for Pregnancy OUD in Jail
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00381845; 1R34DA056014-01A1 (NIH)
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Jail staff at pilot jails (Experimental): Jail staff will be asked to use the implementation resource with guided facilitation to care for pregnant people in and leaving custody.
  Interventions: Other: Maternal Opioid use Disorder Management and Care Resources (MOM CARE) in Custody

INTERVENTIONS:
Other: Maternal Opioid use Disorder Management and Care Resources (MOM CARE) in Custody — MOM CARE is a web-based implementation resource designed for jail staff to help the staff provide evidence-based, trauma-informed and patient-centered care and support to pregnant people with opioid use disorder in and leaving custody. MOM CARE's content will include medical guidance and best-practices from intake to discharge, reentry steps and recommendations, and implementation 'how to' content. There will be specific content for jail administrators, medical and custody staff. Content will be curated from existing resources regarding this topic with new original tools specific to pregnant people with OUD in jail.

SUMMARY:
The goal of this clinical trial is to pilot an adaptable, user-friendly, web-accessible toolkit and implementation strategy for jails to be able to provide access to pregnancy-specific opioid use disorder (OUD) care. The main question it aims to answer is:

- What support and tools do jails that vary in size, resources, and health care delivery systems need for pregnancy care that can be tailored to the environment?

Jail staff will use the implementation resource to provide care to pregnant people in and leaving custody through facilitated guidance. While using the resource, jail staff will:

* Complete 6-month and 12-month surveys assessing the participants use of the tool
* Complete baseline, 6-month, and 12-month qualitative interviews assessing the participants perspectives on using the tool
* Report de-identified jail outcomes data monthly on the pregnant people in the jail's care
* Report jail policy and financial data as it pertains to pregnant people with OUD at baseline Pregnant people with OUD in custody at pilot jails will be asked to participate in qualitative interviews as baseline and 1- and 6 months after release to assess the participants perspectives on the care received in jail and continuity of care.

DETAILED DESCRIPTION:
Ensuring jails provide access to medications for opioid use disorder (MOUD), and in ways that are tailored to the distinctive medical, mental health and social structural aspects of care for pregnant people with OUD is essential for improving short and long-term pregnancy, recovery, and intergenerational outcomes. This project will engage multiple stakeholders, including directly impacted people, to design then pilot a patient-centered and jail-feasible implementation strategy that will facilitate and enhance jails' implementation of MOUD for pregnant people. The strategy will contain a menu of tools to assist jails with immediate needs to provide MOUD to pregnant people entering jails; with pregnancy-tailored counseling; and with other support services and linkages to care that center the obstetrical, psychosocial, and structural needs of this population. The implementation strategy will also be adaptable to a variety of types and geographies of jails. The strategies will then be piloted at four jails with different baseline capacities and services for MOUD for pregnant people.

Study Design. The investigators will conduct this pilot study to assess feasibility of facilitation of use of a web-based resource bundle to help jail workers be able to implement programs and provide care for pregnant people with OUD (PPwOUD). The investigators will design the bundle and then the research team will train jail staff (clinicians and administrators) at 4 pilot sites on how to use each element of the website-- where things are, and how to adapt it to the local environment. The investigators will then measure implementation outcomes at the jail with staff and with implementing care practices, as well as patient level outcomes.

The investigators will do the pilot sequentially, starting with two jails in cohort A and then, six months later, the two jails in cohort B.The investigators will follow the same procedures at each pair of sites

Pilot sites and champions. The investigators will pilot the resource package at jails with combinations of different geography and availability of MOUD for pregnant people. These strata allows for testing and refinement of the bundle tools to be useful to jails with differing local resources, differing frequencies of encountering pregnant people, and differing stages of providing MOUD for pregnant people. While 3 sites provide MOUD in some capacity in pregnancy, all have self-identified needs for enhancements due to lack of pregnancy specificity and numerous challenges in the care for pregnant people with opioid use disorder (PPwOUD). Pilot site #4, with no MOUD will be recruited through existing networks and, as outlined in support letters, with assistance of Sheriffs from confirmed pilot sites. Each jail will identify 1-2 champions for the implementation effort (e.g. nurse, clinician, social worker, health admin).

Facilitated delivery of the bundle. The implementation strategy of facilitation provides human support to promote self-efficacy, persistence, and problem solving; it is rooted in the notion that implementation is a social activity that reflects interpersonal relationships, learning, and people's decisions in a relational context. The team will adapt the integrated Promoting Action on Research Implementation in Health Services (i-PARIHS) facilitation checklist with a blended approach that includes external and internal facilitation. At baseline, the team will conduct in-person or video conference sessions (dependent on jail location) to orient pilot site champions, jail staff and key community partners to the implementation strategy and bundle, followed by monthly video-conference check-ins. Modeling after the Network for the Improvement of Addiction Treatment (NIATx) process improvement model currently being tested at 48 jails. The investigators will deliver well-structured mentoring and technical assistance to jails as to use the bundle to improve care and coordination for pregnant people with OUD. NIATx is an organizational change approach that aims to gauge performance and improve processes by pairing a coach with a site to identify ways to implement change and monitor performance. The investigators will incorporate regularly scheduled outreach to assist, and assess competency of, community partners (e.g. probation, parole, child welfare services, community opioid treatment providers) with justice-involved pregnant populations. The coaching will assist jail leaders and staff to identify local resources, services, agencies, and tools that are relevant for that geographic setting. This focus underlines that toolkits alone have limited impact on implementation outcomes, and successful toolkits benefit from natural internal facilitation.

The intervention is exposing jail staff to a web-based resource that the investigators will design for this study that contains practical, evidence based information on clinical best practices adapted to jail settings for providing medications for OUD for pregnant women in custody AND that contains an implementation strategy for leaders to be able to implement programs.

ELIGIBILITY:
Jail staff Inclusion:

* Jail custody staff who are employed at a jail that holds pregnant women with OUD and are involved in the care of pregnant women with opioid use disorder

Exclusion:

* non-English speaking

Pregnant people with opioid use disorder Inclusion:

* pregnant people with OUD who are in custody at a pilot jail during the study period
* jail stay of at least 24 hours

Exclusion:

* non-English speaking
* women who are intoxicated or actively withdrawing
* women are actively psychotic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2026-01-21 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in organizational readiness as assessed by the ORIC scale | Baseline, 6 months, 12 months
  Staff surveys will be administered to assess organizational readiness at baseline before implementation using the organizational readiness for implementing change (ORIC) scale. The scale is a 12-item instrument used to assess how staff at an organization feel they can implement the change in process proposed by an intervention. Each instrument item uses a Likert scale from 1 (disagree) to 5 (agree). A higher score indicates higher organizational readiness.
Change in technology usage, attitudes and satisfaction as assessed by the UTAUT | 6 months, 12 months
  Staff interviews will be administered to assess technology usage, attitudes and satisfaction using the unified theory of acceptance and use of technology (UTAUT). The UTAUT uses four constructs to determine user acceptance and usage behavior that include performance expectancy, effort expectancy, social influence and facilitating conditions. UTAUT proposes sub-constructs for each of the 4 categories that we will use to inform the interview guide.
Satisfaction, autonomy, discrimination and other experiences for pregnant people with OUD (PPwOUD) in jail as assessed by the RRDS | Post release from jail up to 1 month
  Mixed methods will be used to assess patient-level outcomes for PPwOUD who are in each jail during the pilot phase. Collecting both quantitative and qualitative data that can be triangulated is necessary to assess health outcomes and experiential dimensions of how the jail's bundle implementation affects patient care in and out of jail. The Recovery-related Discrimination Scale (RRDS) is designed to assess self-reported perceived frequency of personal experiences of slights and violation of personal rights due to their alcohol or drug problems. It includes micro and macro discrimination items that are scored from 'never' to 'often.' The more often the items occurred, the more discrimination the individual experienced. These scale questions will inform the interview guide.

SECONDARY OUTCOMES:
Change in financial assessment of caring for PPwOUD in jail | Baseline, 12 months
  The pilot jail budget reports on costs associated with MOUD care in pregnancy will be used to assess any change between baseline and 12 months.
Change in relational coordination as assessed by the Relational Coordination Survey | baseline, 6 months, 12 months
  Staff surveys will be administered at baseline, before implementation, to assess relational coordination using the Relational Coordination (RC) Survey. The survey is a seven-question instrument based on the theory of relational coordination used to assess the impact of relational coordination between staff on desired performance outcomes and assess the impact of individual, organizational, and contextual factors. Jail staff participants will fill this out at baseline, midpoint, and endpoint. Instrument uses a Likert scale from 1 to 5. Scores range from a minimum of 7 to a maximum of 35, with higher scores indicating greater coordination. The results can be calculated as a single Relational Coordination (RC) Index by averaging the responses to all seven questions, or by analyzing scores for each dimension separately.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Sufrin, MD, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Wicomico County Corrections Center, Salisbury, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vilsaint CL, Hoffman LA, Kelly JF. Perceived discrimination in addiction recovery: Assessing the prevalence, nature, and correlates using a novel measure in a U.S. National sample. Drug Alcohol Depend. 2020 Jan 1;206:107667. doi: 10.1016/j.drugalcdep.2019.107667. Epub 2019 Oct 25. PMID 31780300
- [Background] Connolly SL, Sullivan JL, Ritchie MJ, Kim B, Miller CJ, Bauer MS. External facilitators' perceptions of internal facilitation skills during implementation of collaborative care for mental health teams: a qualitative analysis informed by the i-PARIHS framework. BMC Health Serv Res. 2020 Mar 4;20(1):165. doi: 10.1186/s12913-020-5011-3. PMID 32131824
- [Background] Hunter SC, Kim B, Mudge A, Hall L, Young A, McRae P, Kitson AL. Experiences of using the i-PARIHS framework: a co-designed case study of four multi-site implementation projects. BMC Health Serv Res. 2020 Jun 23;20(1):573. doi: 10.1186/s12913-020-05354-8. PMID 32576197
- [Background] Shea CM, Jacobs SR, Esserman DA, Bruce K, Weiner BJ. Organizational readiness for implementing change: a psychometric assessment of a new measure. Implement Sci. 2014 Jan 10;9:7. doi: 10.1186/1748-5908-9-7. PMID 24410955
- [Background] Molfenter T, Vechinski J, Taxman FS, Breno AJ, Shaw CC, Perez HA. Fostering MOUD use in justice populations: Assessing the comparative effectiveness of two favored implementation strategies to increase MOUD use. J Subst Abuse Treat. 2021 Sep;128:108370. doi: 10.1016/j.jsat.2021.108370. Epub 2021 Mar 17. PMID 33762145